CLINICAL TRIAL: NCT07198893
Title: Pattern and Impact of Prehospital Stroke Care on Patient Outcome: A Population-Based Study
Brief Title: Impact of Prehospital Stroke Care Patterns on Clinical Outcomes in Acute Stroke Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Refat Hamed Khalaf Ahmed, resident at the Neuropsychiatry department, Assiut University
Other Study IDs: Prehospital Stroke Care
Record Dates: First submitted 2025-09-20; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Prehospital Stroke Care
Keywords: Prehospital Stroke Care; Patient Outcome:

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adults who present with acute stroke: The study population consists of adults who present with acute stroke and have sought or received prehospital care within the hospital's catchment area. Participants are adult patients aged 18 years and above with an acute ischemic or hemorrhagic stroke diagnosis confirmed by neuroimaging

SUMMARY:
This study evaluates how prehospital care factors, including stroke awareness, emergency response, transport, and referral processes, impact patient outcomes in acute stroke cases.

DETAILED DESCRIPTION:
The research is a population-based observational cohort study conducted at Assiut University Hospital's Neuropsychiatry Department. It investigates patterns of prehospital stroke care with a focus on patient and caregiver awareness of stroke symptoms, the type of first medical contact, transport modes, referral pathways, and emergency medical service response. The study aims to understand how these prehospital factors influence stroke outcomes, including timely access to treatment, functional recovery, and mortality rates. Standardized tools, structured questionnaires, EMS records, and hospital medical data will be used to collect comprehensive information.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age

Confirmed diagnosis of acute stroke (ischemic/hemorrhagic) verified by CT or MRI

Residents of the study's defined geographical area

Patients who experienced stroke and sought prehospital care pathways (EMS or direct hospital presentation)

Informed consent from the patient or legally authorized representative

Exclusion Criteria:

* Patients with transient ischemic attack (TIA) or stroke mimics without confirmed acute stroke diagnosis

Missing or incomplete data on prehospital care

Patients unable or unwilling to provide consent without a representative available

Non-residents or visitors outside the designated geographical area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are adult patients aged 18 years and above with an acute ischemic or hemorrhagic stroke diagnosis confirmed by neuroimaging. All patients must reside within the defined geographical area and have used emergency medical services or presented directly with stroke symptoms. Caregivers will also provide data regarding symptom recognition and decision-making. Patients with stroke mimics, incomplete records, or without consent will be excluded.
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Stroke symptom awareness | Baseline
  Assessment of general knowledge and recognition of stroke symptoms and prehospital care pathways will be measured using the Stroke Knowledge Test (SKT), a validated questionnaire.
  The SKT consists of 20 multiple-choice questions evaluating recognition of stroke symptoms and knowledge of emergency response. Scores range from 0 to 20, with higher scores indicating greater awareness and better knowledge.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zachrison KS, Nielsen VM, de la Ossa NP, Madsen TE, Cash RE, Crowe RP, Odom EC, Jauch EC, Adeoye OM, Richards CT. Prehospital Stroke Care Part 1: Emergency Medical Services and the Stroke Systems of Care. Stroke. 2023 Apr;54(4):1138-1147. doi: 10.1161/STROKEAHA.122.039586. Epub 2022 Nov 29. PMID 36444720